CLINICAL TRIAL: NCT00522145
Title: A Phase 2 Study of XL647 in Subjects With Non-Small Cell Lung Cancer Who Have Progressed After Responding to Treatment With Either Gefitinib or Erlotinib
Brief Title: Study of XL647 in Subjects With NSCLC Who Have Progressed After Responding to Treatment With Gefitinib or Erlotinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL647-203
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — XL647

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group 1 (Experimental)
  Interventions: Drug: XL647

INTERVENTIONS:
Drug: XL647 — Daily dosing as a single oral agent at a dose of 300 mg supplied as 50-mg tablets
  Other Names: KD019

SUMMARY:
The purpose of this study is to determine the best confirmed response rate of daily administration of the multiple receptor tyrosine kinase (RTK) inhibitor (including EGFR and VEGFR2) XL647 in subjects with NSCLC who have progressed after responding to treatment with either erlotinib or gefitinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of unresectable Stage IIIB or Stage IV relapsed or recurrent NSCLC.
* Subjects must have:

  1. documented (radiological or clinical) progressive disease (PD) following a prior response (including stable disease) to monotherapy with erlotinib or gefitinib that was administered for at least 12 weeks prior to progression OR
  2. a documented T790M EGFR mutation
* Measurable disease defined according to RECIST
* ECOG performance status of 0 or 1.
* Sexually active subjects must use an accepted method of contraception during the course of the study.
* Female subjects of childbearing potential must have a negative pregnancy test at enrollment.

Exclusion Criteria:

* Received radiation to ≥25% of his or her bone marrow within 30 days of XL647 treatment.
* Received erlotinib or gefitinib, or other anticancer therapy within 14 days of the first dose of study drug.
* Received an investigational drug (excluding erlotinib or gefitinib) within 30 days of the first dose of study drug.
* Receiving anticoagulation therapy with warfarin.
* Not recovered to Grade ≤1 from adverse events (AEs) due to antineoplastic agents, investigational drugs, or other medications that were administered prior to study enrollment.
* Corrected QT interval (QTc) of >0.45 seconds.
* Progressive, symptomatic, or hemorrhagic brain or leptomeningeal metastases.
* Requires steroid or anticonvulsant therapy for the treatment of brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Determine the best confirmed response rate | Inclusion until disease progression

SECONDARY OUTCOMES:
Safety and tolerability of XL647 administered daily | First treatment until 30 day post last treatment
Progression-free survival, duration of response, and overall survival | Incusion until disease progression
Further characterize the pharmacokinetic (PK) parameters | Every 8 weeks after Day 57 until disease progression

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Ronald Yanagihara, Gilroy, California
  - University of California Davis Cancer Center, Sacramento, California
  - Oncology Division and General Clincial Research, Stanford University Medical Center, Stanford, California
  - Cancer Care Center, Inc. P.C., New Albany, Indiana
  - Washington County Hospital, The Center for Clinical Research, Hagerstown, Maryland
  - Wayne State University, Wertz Clinical Cancer Center, Karmanos Center, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New Bern Cancer Care Oncology, New Bern, North Carolina
  - Case Western Reserve University, University Hospitals of Cleveland, Cleveland, Ohio
  - Signal Point Clinical Research Center, Middletown, Ohio

REFERENCES:
- [Background] Pietanza MC, Lynch TJ Jr, Lara PN Jr, Cho J, Yanagihara RH, Vrindavanam N, Chowhan NM, Gadgeel SM, Pennell NA, Funke R, Mitchell B, Wakelee HA, Miller VA. XL647--a multitargeted tyrosine kinase inhibitor: results of a phase II study in subjects with non-small cell lung cancer who have progressed after responding to treatment with either gefitinib or erlotinib. J Thorac Oncol. 2012 Jan;7(1):219-26. doi: 10.1097/JTO.0b013e31822eebf9. PMID 22011666